CLINICAL TRIAL: NCT05505448
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled Study to Assess the Safety, Tolerability, Pharmacokinetics, and Immunogenicity of a Regeneron Anti-SARS-CoV-2 Monoclonal Antibody (a COVID-19 Therapeutic) in Adult Healthy Volunteers
Brief Title: A Trial to Learn if a COVID-19 Therapeutic is Safe and Well Tolerated, and How it Works in the Body of Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R14284-HV-2253; 2022-002181-33 (EudraCT Number)
Record Dates: First submitted 2022-08-15; First posted 2022-08-17 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Healthy
Keywords: Coronavirus disease 2019 (COVID-19) vaccinated; Negative SARS-CoV-2 diagnostic test within approximately ≤72 hours of randomization
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Cohort 1 Mid IV Dose (Experimental): Randomized 3:1 for single ascending dose
  Interventions: Drug: REGN14284; Drug: Matching Placebo
- Cohort 2 Mid SC Dose (Experimental): Randomized 3:1 for single ascending dose
  Interventions: Drug: REGN14284; Drug: Matching Placebo
- Cohort 3 High IV Dose (Experimental): Randomized 3:1 for single ascending dose
  Interventions: Drug: REGN14284; Drug: Matching Placebo
- Cohort 4 High SC Dose (Experimental): Randomized 3:1 for single ascending dose
  Interventions: Drug: REGN14284; Drug: Matching Placebo
- Cohort 5 Higher IV Dose (Experimental): Randomized 3:1 for single ascending dose
  Interventions: Drug: REGN14284; Drug: Matching Placebo
- Cohort 6 Highest IV Dose (Experimental): Randomized 3:1 for single ascending dose
  Interventions: Drug: REGN14284; Drug: Matching Placebo
- Cohort 7 Low IV Dose (Experimental): Randomized 3:1 for single ascending dose
  Interventions: Drug: REGN14284; Drug: Matching Placebo
- Cohort 8 Low SC Dose (Experimental): Randomized 3:1 for single ascending dose
  Interventions: Drug: REGN14284; Drug: Matching Placebo

INTERVENTIONS:
Drug: REGN14284 — Single ascending intravenous (IV) or subcutaneous (SC) administration per the protocol
Drug: Matching Placebo — Single ascending IV or SC administration per the protocol

SUMMARY:
The primary objective of the study is to evaluate the safety and tolerability of REGN14284 in healthy participants, as measured by all treatment-emergent adverse events (TEAEs) and treatment-emergent serious adverse events (SAEs).

The secondary objectives of the study are:

* To assess the concentration-time profile of REGN14284 in serum
* To assess the immunogenicity of REGN14284

ELIGIBILITY:
Key Inclusion Criteria:

1. Has SARS-CoV-2-negative test result from a sample collected ≤72 hours prior to randomization as described in the protocol.
2. Has received complete primary series of standard-of-care COVID-19 vaccination per local guidance, completed at least 2 weeks prior to screening
3. Has a body mass index (BMI) between 18 and 31 kg/m2 (inclusive) at the screening visit
4. Is judged by the investigator to be in good health based on medical history, physical examination, vital sign measurements, laboratory safety testing and ECGs performed at screening and/or prior to administration of study drug

Key Exclusion Criteria:

1. History of clinically significant cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, infectious, autoimmune, oncologic, psychiatric or neurological disease, as assessed by the investigator as described in the protocol
2. Presents any concern to the investigator that might confound the results of the study or poses an additional risk to the participant by their participation in the study
3. Was hospitalized (ie, >24 hours) for any reason within 30 days of the screening visit
4. Has a history of alcohol or drug abuse as determined by the investigator
5. Has a history of significant multiple and/or severe allergies, or has had an anaphylactic reaction to drugs or food as described in the protocol
6. Use of any medications or nutritional supplements within approximately 5 half-lives or 2 weeks, whichever is longer, prior to first administration of the study drug through the end of the study, except for the permitted medications listed as described in the protocol
7. Participated in any clinical research study evaluating another investigational drug including biologics or specific immunotherapy, within at least 5 half-lives or 90 days (whichever is longer) of an investigational biologic drug, or at least 4 weeks for small molecules or other investigational drugs, prior to the screening visit

NOTE: Other protocol defined inclusion / exclusion criteria apply

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Occurrence and severity of all treatment emergent adverse events (TEAEs) | Through approximately day 169
Occurrence and severity of all severe adverse events (SAEs) | Through approximately day 169

SECONDARY OUTCOMES:
Concentrations of REGN14284 in serum over time | Through approximately day 169
Incidence of Anti-drug antibodies (ADAs) to REGN14284 over time | Through approximately day 90
Titer of ADAs to REGN14284 over time | Through approximately day 90

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (1):
- Universitair Ziekenhuis Leuven Gasthuisberg Campus, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication, has made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry), has the legal authority to share the data, and has ensured the ability to protect participant privacy.
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/